CLINICAL TRIAL: NCT06755437
Title: Self Treatment With an Electronic Device for Cognitive Rehabilitation in Patients With Subacute Stroke: A Randomized Controlled Trial
Brief Title: Self Treatment With an Electronic Device for Cognitive Rehabilitation in Patients With Subacute Stroke
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated early due to recruitment challenges related to the large sample size required to achieve adequate statistical power.
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Valentina Varalta, Doctor, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 269666
Record Dates: First submitted 2024-12-18; First posted 2025-01-01 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2024-10

CONDITIONS: Stroke; Cognitive Deficits; Computerized Rehabilitation; Computerized Device
Keywords: stroke; neuropsychological rehabilitation
MeSH Terms: conditions — Stroke; Cognition Disorders | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rehabilitation with a computerized device (Experimental): Every morning both groups received the same face-to-face cognitive treatment using an electronic device. in the afternoon only the experimental group performed self-treatment with the same device for 2 weeks, 5 sessions a week, for a total of 10 sessions.
  Interventions: Device: Rehabilitation with a computerized device (in the morning); Device: Self-treatment with a computerized device (in the afternoon)
- Rehabilitation with pencil-and-paper exercises (Active Comparator): Every morning both groups received the same face-to-face cognitive treatment using an electronic device. Only the control group performed self-treatment with paper-and-pencil exercises for 2 weeks, 5 sessions a week, for a total of 10 sessions.

INTERVENTIONS:
Device: Rehabilitation with a computerized device (in the morning) — Each group received face-to-face cognitive rehabilitation with the electronic device for 45 min. The exercises were selected by the therapist and divided into four sessions of 2 to 3 days each. Each session included 40 min of activity and 5 minute of break
  Arms: Rehabilitation with a computerized device
Device: Self-treatment with a computerized device (in the afternoon) — In the afternoon, the experimental group performed 60 min. self-guided treatment with the electronic device.
  Arms: Rehabilitation with a computerized device
Behavioral: self-treatment with pencil-and-paper exercises (in the afternoon) — In the afternoon, the control group performed 60 min of cognitive self-treatment with conventional paper-and-pencil instruments. The therapist created a variety of exercises every day

SUMMARY:
The objective of this study is to evaluate whether the independent use of an electronic device by a patient with stroke outcomes can enhance the effectiveness of rehabilitative treatment for attentional functions compared to standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ischemic or hemorrhagic stroke
* Within 2 weeks since stroke onset
* Age under 85 years
* Attention deficits as measured by the Trails task or the Broken Hearts subtest in the Oxford Cognitive Screen (OCS)

Exclusion criteria:

* Visual impairment documented by clinical history (e.g., cataracts, diabetic retinopathy, glaucoma, hemianopia)
* Uncompensated psychiatric disorders
* Drug or alcohol abuse
* History of dementia
* Severe comprehension disorders as determined by the Semantics subtest in the Oxford Cognitive Screen (OCS)
* Spatial neglect as determined by the Broken Hearts subtest in the OCS

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Trail Making Test Part A (TMT-A) | From enrollment (within 2 weeks of stroke onset) to the completion of treatment (2 weeks after the start of treatment)
  The Trail Making Test Part A (TMT-A) is a neuropsychological assessment that measures selective attention and processing speed. Participants connect a series of numbered circles in sequential order as quickly as possible. The score is determined by the time taken to complete the task, with shorter times indicating better performance. Errors may negatively impact the score.

SECONDARY OUTCOMES:
Trail Making Test Part B (TMT-B) | From enrollment (within 2 weeks of stroke onset) to the completion of treatment (2 weeks after the start of treatment)
  The Trail Making Test Part B (TMT-B) is a neuropsychological test that measures Divided attention. Participants must connect numbered and lettered circles in alternating order as quickly as possible. The score is based on the time taken to complete the test, with shorter times indicating better performance. Any errors may negatively impact the score.
Dual task test | From enrollment (within 2 weeks of stroke onset) to the completion of treatment (2 weeks after the start of treatment)
  Dual Task to assess the ability to perform two tasks simultaneously (one verbal and one visuomotor). Performance is evaluated based on accuracy and speed in both tasks, providing insight into how well an individual can manage competing cognitive and motor demands.
short version of the Elithorn's Perceptual Maze Test | From enrollment (within 2 weeks of stroke onset) to the completion of treatment (2 weeks after the start of treatment)
  The short version of the Elithorn's Perceptual Maze Test has a score range from 0 to 16, where the score is determined by the number of errors made during the task. Fewer errors correspond to better performance, with 0 indicating no errors and 16 representing the maximum number of errors. This test assesses planning, attention, and problem-solving skills, with lower scores reflecting more efficient cognitive functioning.
Stroop Test | From enrollment (within 2 weeks of stroke onset) to the completion of treatment (2 weeks after the start of treatment)
  The Stroop Test is a neuropsychological tool that assesses cognitive flexibility, selective attention, and the ability to inhibit automatic responses. Participants are required to name the color of the ink in which a word is printed, rather than reading the word itself. The score is based on the time taken to complete the task and the number of errors made when naming the ink colors. A higher score indicates more errors or a slower completion time, reflecting challenges in cognitive control and attention.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Universitaria Integrata Verona - UOC di Neuroriabilitazione, Verona, Italy